CLINICAL TRIAL: NCT02017743
Title: Effectiveness And Safety of LMWH Treatment in Cancer Patients Diagnosed With Non-High Risk Venous Thromboembolism - An Observational Study
Brief Title: Effectiveness And Safety of LMWH Treatment in Cancer Patients Diagnosed With Non-High Risk Venous Thromboembolism
Acronym: TREBECA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Trio Grup Clinical Research (Industry)
Responsible Party: Sponsor
Other Study IDs: TREBECA
Record Dates: First submitted 2013-12-05; First posted 2013-12-23 (Estimated); Last update posted 2013-12-23 (Estimated); Status verified 2013-12

CONDITIONS: Venous Thromboembolism
MeSH Terms: conditions — Venous Thromboembolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study is a multicenter post authorization observational study. Cancer patients diagnosed with non high risk VTE and are followed up in an outpatient setting will be treated with LMWH and the data will be recorded. Since this is an observational study there are no specific treatment protocols, i.e., patients will be treated according to the best investigator's criteria. Treatment protocol will be based on the routine treatment practice of the involved investigator. Patients to enroll will be cancer patients diagnosed for VTE and who are able to receive outpatient LMWH treatment. There will be no specific hypothesis to be tested.

DETAILED DESCRIPTION:
Inclusion criteria

* 18 years or upper age
* A signed informed consent document
* Cancer patient diagnosed for VTE
* Life expectancy > 6 months
* Eligible for criteria of outpatient administration of LMWH

Exclusion criteria

• Should not carry any medical situation listed below, that outpatient administration of LMWH might be risky :

1. Patients with active bleeding or at-risk for bleeding
2. Major surgery in the last 7 days
3. Cardiopulmonary unstability
4. Severe systemic venous occlusion
5. Patients at high risk for pulmonary embolism
6. Thrombocytopenia (<50000/microliter)
7. Inpatients under medical or surgery supervision
8. Patients with low ability to communicate and for whom it is not possible to provide care at home
9. INR≥1.5 due to liver functions impairment
10. Diagnosed for cerebral vascular aneurism
11. Active gastric and/or duodenum ulcer
12. Diagnosed for bacterial endocarditis
13. Severe renal function impairment (Creatinine clearance < 30 ml/min)
14. Grade 3 hypertension (DBP >= 110 mmHg and/or SBP >= 180 mmHg)
15. <35 kg or ≥110 kg weight
16. Known allergy to heparin and/or its derivatives
17. History of cerebrovascular event in the last 1 month
18. Active haemorrhage within the last 3 months

ELIGIBILITY:
Inclusion Criteria:

* 18 years or upper age
* A signed informed consent document
* Cancer patient diagnosed for VTE
* Life expectancy > 6 months
* Eligible for criteria of outpatient administration of LMWH

Exclusion Criteria:

* Patients with active bleeding or at-risk for bleeding
* Major surgery in the last 7 days
* Cardiopulmonary unstability
* Severe systemic venous occlusion
* Patients at high risk for pulmonary embolism
* Thrombocytopenia (<50000/microliter)
* Inpatients under medical or surgery supervision
* Patients with low ability to communicate and for whom it is not possible to provide care at home
* INR≥1.5 due to liver functions impairment
* Diagnosed for cerebral vascular aneurism
* Active gastric and/or duodenum ulcer
* Diagnosed for bacterial endocarditis
* Severe renal function impairment (Creatinine clearance < 30 ml/min)
* Grade 3 hypertension (DBP >= 110 mmHg and/or SBP >= 180 mmHg)
* <35 kg or ≥110 kg weight
* Known allergy to heparin and/or its derivatives
* History of cerebrovascular event in the last 1 month
* Active haemorrhage within the last 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients to enroll will be cancer patients diagnosed for VTE and who are able to receive outpatient LMWH treatment.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2012-12; Primary Completion 2014-08 (Estimated); Study Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
Evaluation of effectiveness of LMWH used in the treatment of thrombosis in cancer patients with VTE regarding new thrombosis. | [Time to new thrombosis in 15 days]
Evaluation of effectiveness of LMWH used in the treatment of thrombosis in cancer patients with VTE regarding resolution. | [Time to resolution in 15 days]
Evaluation of effectiveness of LMWH used in the treatment of thrombosis in cancer patients with VTE regarding bleeding | [Time to bleeding in 15 days]

CONTACTS AND LOCATIONS:
Overall Officials: Metin Ozkan, Prof., Principal Investigator — Erciyes University Faculty of Medicine
Locations (1):
- Erciyes University Faculty of Medicine, Kayseri, Melikgazi, Turkey (Türkiye)